CLINICAL TRIAL: NCT05923489
Title: Routine Angiography Follow-Up After Percutaneous Coronary Intervention in High-Risk Patients (The REVISE Trial)
Brief Title: Routine Angiography Follow-Up After Percutaneous Coronary Intervention in High-Risk Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Jinhua Central Hospital (Other); Changxing People's Hospital (Other); The Affiliated Hospital of Hangzhou Normal University (Other); Second Affiliated Hospital of Shantou University Medical College (Other); Dongyang People's Hospital (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Huizhou Municipal Central Hospital (Other); First Affiliated Hospital of Ningbo University (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-0332
Record Dates: First submitted 2023-06-20; First posted 2023-06-28 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine Angiography Follow-up (RAF) group (Experimental): Patients in the RAF group will have routine angiography follow-up at 12 months after revascularization.
  Interventions: Diagnostic Test: Routine Angiography Follow-up
- Routine Clinical Follow-up (RCF) group (Active Comparator): Patients in the RCF group will have routine clinical follow-up at 12 months after revascularization, and the physician will decide whether further invasive testing is needed.
  Interventions: Diagnostic Test: Routine Clinical Follow-up

INTERVENTIONS:
Diagnostic Test: Routine Angiography Follow-up — Patients in the RAF group will have routine angiography follow-up at 12 months after revascularization.
  Arms: Routine Angiography Follow-up (RAF) group
Diagnostic Test: Routine Clinical Follow-up — Patients in the RCF group will have routine clinical follow-up at 12 months after revascularization, and the physician will decide whether further invasive testing is needed.
  Arms: Routine Clinical Follow-up (RCF) group

SUMMARY:
Comparison of clinical outcomes between routine angiography follow-up and routine clinical follow-up after percutaneous coronary intervention in high-risk patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Successful PCI with at least two of the following high-risk factors:

A. Left main lesion; B. Bifurcation lesion (true bifurcation); C. Ostial lesion of main vessels (left anterior descending, left circumflex artery, right coronary artery); D. Chronic total occlusion; E. Multivessel revascularization (≥ 2 vessels); F. In-stent restenosis; G. Diffuse long lesion (lesion length ≥ 30 mm or stent length ≥ 38 mm); H. Severe calcified lesion (Significant severe calcification on angiography); I. Bypass graft lesion; J. Diabetes mellitus; K. Chronic kidney disease (defined as an estimated glomerular filtration rate of <30 ml per minute per 1.73 m2 of body-surface area or the receipt of dialysis); L. Myocardial infarction;

- He/she or his/her legally authorized representative provides written informed

Exclusion Criteria:

* Revascularization with bare metal stents and/or balloon angioplasty with non-drug-coated balloons.
* Pregnant and/or lactating women.
* Life expectancy of less than 2 years.
* Repeat interventional therapy is planned.
* Subject was unable to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2618 (Estimated)
Dates: Start 2023-10-26 (Actual); Primary Completion 2026-10-15 (Estimated); Study Completion 2029-10-15 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint of all-cause death, myocardial infarction, or hospitalization for unstable angina | 24 months
  The rate of a composite endpoint of all-cause death, myocardial infarction, or hospitalization for unstable angina

SECONDARY OUTCOMES:
Composite endpoint of all-cause death, myocardial infarction, or hospitalization for unstable angina | 60 months
  The rate of a composite endpoint of all-cause death, myocardial infarction, or hospitalization for unstable angina
All-cause death | 24 and 60 months
  The rate of all-cause death
Myocardial infarction | 24 and 60 months
  The rate of myocardial infarction
Hospitalization for unstable angina | 24 and 60 months
  The rate of hospitalization for unstable angina
Cardiac death | 24 and 60 months
  The rate of hospitalization for cardiac death
Invasive angiography during follow-up | 24 and 60 months
  The rate of invasive angiography during follow-up
Any revascularization | 24 and 60 months
  The rate of any revascularization during follow-up (ischemia-driven vs. all-cause)
Revascularization of any target vessel/lesion | 24 and 60 months
  The rate of revascularization of any target vessel/lesion
Revascularization of any non-target vessel/lesion | 24 and 60 months
  The rate of revascularization of any non-target vessel/lesion
Health Economics Analysis (cost-effectiveness) | 24 and 60 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided